CLINICAL TRIAL: NCT05915910
Title: Prospective Collection of Biospecimen in Pediatric Patients and Adult Guardians Diagnosed With Glycogen Storage Disease Type 1B (GSD1b)
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit additional subjects due to disease rarity
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-09747
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Glycogen Storage Disease Type IB
MeSH Terms: conditions — Glycogen Storage Disease IB

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GSD1b G339C Homozygous (n=3)
  Interventions: Diagnostic Test: Specimen Donation
- GSD1b L348FS Homozygous (n=3)
  Interventions: Diagnostic Test: Specimen Donation
- GSD1b G339C/ L348FS Heterozygous (n=3)
  Interventions: Diagnostic Test: Specimen Donation
- GSD1b Parents (n=6)
  Interventions: Diagnostic Test: Specimen Donation

INTERVENTIONS:
Diagnostic Test: Specimen Donation — blood donation

SUMMARY:
The primary objective of this study is to collect whole blood from patients diagnosed with Glycogen storage disease type 1B, which will be used to support the investigation of potential therapies that address the genetic basis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 4-85
* Subjects that are diagnosed with Glycogen Storage Disease Type Ib (GSD1b, von Gierke disease)
* Subjects who are G339C Homozygous or L348FS Homozygous or G339C/ L348FS heterozygous or are the biological parent of subjects diagnosed with Glycogen Storage Disease Type Ib (GSD1b, von Gierke disease) and are a biological parent of a subject in Cohort 1 (G339C homozygous) or Cohort 2 (L348FS homozygous)
* Subjects or guardians must be willing and able to provide appropriate photo identification to mobile phlebotomist during at-home visit for verification of identity
* Subjects and/or Guardians must be willing and able to provide appropriate written informed consent and/or assent, as applicable

Exclusion Criteria:

* Subjects will be excluded if they experienced excess blood loss, including blood donation defined as 250 mL in the last month or 500 mL in the last two months. For subjects in the pediatric population, subjects will be excluded if they experienced excess blood loss, including blood donation defined as 3 mL/kg or up to 50 mL in the last 8-weeks.
* For requests that do not include pregnant subjects, subjects will be excluded if they are pregnant or nursing.
* For requests that do not include subjects with infectious diseases, subjects will be excluded if they have current, active HIV, hepatitis or other infectious diseases (self-reported or medical history reviewed).
* Subjects will be excluded if they have taken an investigational product in the last 30 days.

Ages: 4 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: participants diagnosed with Glycogen storage disease type 1
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Bipspecimen collection from subjects that are diagnosed with Glycogen Storage Disease Type Ib (GSD1b, von Gierke disease); Subjects that are the biological parent of subjects diagnosed with Glycogen Storage Disease Type Ib (GSD1b, von Gierke disease) | 1 Year
  Bipspecimen collection from subjects or their parental guardians that are diagnosed with Glycogen Storage Disease Type Ib(GSD1b, von Gierke disease) for the purpose to analyze the biospecimens to support the investigation of potential therapies that address the genetic basis of this disease. The primary outcome measure is the collection of biospecimens for quantitative analysis using PBMC processes to report cell viability of at least 5M cells per vial.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine BioSciences, Inc., Woburn, Massachusetts, United States